CLINICAL TRIAL: NCT03701516
Title: Clinical Evaluation of Etafilcon A Contact Lenses Using a Novel Molding Process 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6307
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Results first posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TEST/CONTROL (Experimental): Subjects between the ages of 18 and 70 years of age and are habitual wearers of daily disposable contact lens wearers will be randomly assigned to the Test/Control sequence.
  Interventions: Device: etafilcon A with novel molding process; Device: etafilcon A with current molding process
- CONTROL/TEST (Experimental): Subjects between the ages of 18 and 70 years of age and are habitual wearers of daily disposable contact lens wearers will be randomly assigned to the Control/Test sequence.
  Interventions: Device: etafilcon A with novel molding process; Device: etafilcon A with current molding process

INTERVENTIONS:
Device: etafilcon A with novel molding process — TEST Lens
Device: etafilcon A with current molding process — CONTROL Lens

SUMMARY:
This study is a multi-site, group sequential, adaptive, randomized, double-masked, 2×2 crossover design, 1-week dispensing study. Subjects will wear bilaterally both Test and Control lenses in a random order for 1-week each as a daily disposable modality with a wash-out period of 1 week between the wearing periods.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Must be at least 18 and not more than 70 years of age (including 70) at the time of screening.
  4. The subject must be a habitual and adapted wearer of hydrogel daily disposable brand contact lens in both eyes (at least 1 month of daily wear).
  5. The subject must have normal eyes (i.e., no ocular medications or infections of any type).
  6. The subject's required spherical contact lens prescription must be in the range of -1.00 to -4.50 D in each eye.
  7. The subject's refractive cylinder must be < 0.75 D in each eye.
  8. The subject must have best corrected visual acuity of 20/25 or better in each eye.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
  2. Any systemic disease, autoimmune disease, or use of medication that may interfere with contact lens wear.
  3. Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
  4. Any ocular infection.
  5. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
  6. Monovision or multi-focal contact lens correction.
  7. Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
  8. History of binocular vision abnormality or strabismus.
  9. Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g., HIV, by self-report).
  10. Suspicion of or recent history of alcohol or substance abuse.
  11. History of serious mental illness.
  12. History of seizures.
  13. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician)
  14. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion.
  15. Any Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the FDA classification scale.
  16. Any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - EyeCenter Optometrics, Rocklin, California
  - Fleming Island Vision Center, Fleming Island, Florida
  - Bartram Eye Clinic, Jacksonville, Florida
  - Sabal Eye Care, Longwood, Florida
  - Maitland Vision Center, Maitland, Florida
  - St. Johns Eye Associates, Saint Augustine, Florida
  - Sacco Eye Group, Vestal, New York
  - ProCare Vision Centers, Granville, Ohio
  - Eyecare Professionals of Powell, Powell, Ohio
  - Primary Eyecare Group, Brentwood, Tennessee
  - Total Eye Care, PA, Memphis, Tennessee
  - Boutetourt Eyecare, LLC, Salem, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 268 subjects were enrolled in this study. Of those enrolled, 263 dispensed at least one study lens while, 5 subjects failed to meet all eligibility criteria. Of those dispensed subjects, 252 subjects completed the study while, 11 subjects were discontinued from the study.
Groups:
- Test/Control: Subjects randomized to receive the Test lens during the first period and then receive the Control lens during the second period.
- Control/Test: Subjects randomized to receive the Control lens during the first period and then receive the Test lens during the second period.
Period: Period 1
Arm/Group | Test/Control | Control/Test
Started | 131 | 132
Completed | 127 | 127
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 0 | 2
Not completed — Unsatisfactory Lens Fitting due to Test Article | 2 | 0
Not completed — Non Compliance to Protocol | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2
Arm/Group | Test/Control | Control/Test
Started | 127 | 127
Completed | 126 | 126
Not Completed | 1 | 1
Not completed — failed to meet all eligibility creiteria | 1 | 0
Not completed — Unsatisfactory Lens Fitting due to Test Article | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects dispensed in a study lens.
Groups:
- Dispensed Subject: All subjects dispensed a study lens.
Arm/Group | Dispensed Subject
Number analyzed (Participants) | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 186
  Male | 77
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 13
  Black or African American | 17
  White | 228
  Other | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 263

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort Scores
Description: Overall comfort was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 1-week Follow-up
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: unit on a scale
Groups:
- Test: Subjects that wore the Test lens in either the first or second period of the study.
- Control: Subjects that wore the Control lens in either the first or second period of the study.
Arm/Group | Test | Control
Number analyzed (Participants) | 237 | 237
unit on a scale | 59.9 (24.21) | 60.8 (24.69)
Statistical Analysis 1: Comparison: Test vs Control; Test type: Non-Inferiority — Non-inferiority will be established if the lower bound of the credible interval of the mean difference between Test and Control is greater than -5; Bayesian repeated measurement model; Results were reported as regression coefficient mean estimates with credible intervals (CrI); Posterior Mean Difference = -0.38, 98% CI 2-sided [-4.53 to 3.85], Standard Deviation 1.781 — Mean difference was calculated as Test - Control

2. Primary Outcome: Overall Vision Scores
Description: Overall vision was assessed using the CLUE questionnaire. CLUE is a validated PRO questionnaire to assess patient experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using IRT follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 1-week Follow-up
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Test | Control
Number analyzed (Participants) | 237 | 237
unit on a scale | 64.2 (20.06) | 66.5 (19.94)
Statistical Analysis 1: Comparison: Test vs Control; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Bayesian repeated measurement model; Results were reported as regression coefficient mean estimates with credible intervals (CrI); Posterior Mean Difference = -2.34, 98% CI 2-sided [-5.36 to 0.61], Standard Deviation 1.263 — Mean difference was calculated as Test - Control

3. Secondary Outcome: Average Daily Wear Time
Description: Average daily wear time was calculated as the number of hours between subjects reported time of insertion and time of removal of the study lenses, on an average day, at 1-week follow-up evaluation. Higher wear times indicate better lens performance. The average wear time was reported for each lens type.
Time Frame: 1-week Follow-up
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Test | Control
Number analyzed (Participants) | 237 | 237
Hours | 14.3 (1.92) | 14.4 (1.82)
Statistical Analysis 1: Comparison: Test vs Control; Test type: Non-Inferiority — Non-inferiority will be established if the lower bound of the credible interval of the mean difference between Test and Control is greater than -1; Bayesian repeated measurement model; Results were reported as regression coefficient mean estimates with credible intervals (CrI); Posterior Mean Difference = -0.06, 95% CI 2-sided [-0.22 to 0.10], Standard Deviation 0.083 — Mean difference was calculated as Test - Control

4. Secondary Outcome: LLHC LogMAR Visual Performance
Description: Visual performance was calculated as monocular contact lens-corrected distance visual acuity using a logMAR visual acuity scale. This was evaluated under low luminance and high contrast conditions (LLHC) at 4 meters from Early Treatment Diabetic Retinopathy Study (ETDRS) charts at the 1-week follow-up visit. Lower visual performance values indicate better vision. Two measurements were performed for each eye at 1-week follow-up. The average visual performance was reported for each lens type.
Time Frame: 1-week Follow-up
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Test | Control
Number analyzed (Participants) | 237 | 237
Number analyzed (eyes) | 474 | 474
logMAR | -0.059 (0.1123) | -0.060 (0.1176)
Statistical Analysis 1: Comparison: Test vs Control; Test type: Non-Inferiority — Non-inferiority will be established if the upper bound of the credible interval of the mean difference between Test and Control is less than 0.05; Bayesian repeated measurement random-eff; Results were reported as regression coefficient mean estimates with credible intervals (CrI); Posterior Mean Difference = 0.001, 95% CI 2-sided [-0.005 to 0.006], Standard Deviation 0.0028 — Mean difference was calculated as Test - Control

5. Secondary Outcome: HLLC LogMAR Visual Performance
Description: Visual performance was calculated as monocular contact lens-corrected distance visual acuity using a logMAR visual acuity scale. This was evaluated under high luminance and low contrast conditions (HLLC) at 4 meters from Early Treatment Diabetic Retinopathy Study (ETDRS) charts at the 1-week follow-up visit. Lower visual performance values indicate better vision. Two measurements were performed for each eye at 1-week follow-up. The average visual performance was reported for each lens type.
Time Frame: 1-week Follow-up
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Test | Control
Number analyzed (Participants) | 237 | 237
Number analyzed (eyes) | 474 | 474
logMAR | 0.062 (0.1209) | 0.065 (0.1176)
Statistical Analysis 1: Comparison: Test vs Control; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; Bayesian repeated measurement model; Results were reported as regression coefficient mean estimates with credible intervals (CrI); Posterior Mean Difference = -0.003, 95% CI 2-sided [-0.009 to 0.002], Standard Deviation 0.0029 — Mean difference was calculated as Test - Control

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study, approximately 2 weeks per subject.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/263 | 0/263
Serious Adverse Events (participants affected / at risk) | 0/263 | 0/263
Other Adverse Events (participants affected / at risk) | 0/263 | 0/263

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/16/NCT03701516/Prot_SAP_000.pdf